CLINICAL TRIAL: NCT02192294
Title: An Open-label, Randomized, 2-period Crossover Study To Evaluate Absolute Bioavailability Of Bosutinib In Healthy Subjects
Brief Title: Absolute Bioavailability Of Bosutinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1871044; 2014-001405-40 (EudraCT Number)
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Bosutinib; absolute bioavailability
MeSH Terms: interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bosutinib (Experimental)
  Interventions: Drug: Oral Bosutinib; Drug: Intravenous infusion of bosutinib

INTERVENTIONS:
Drug: Oral Bosutinib — a single dose of 500 mg oral bosutinib
Drug: Intravenous infusion of bosutinib — a single dose of 120 mg of bosutinib intravenous infusion (1 hour)

SUMMARY:
This is an open-label, randomized, single-dose, one-cohort, two-sequence, two-period crossover study in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects (of non-childbearing potential).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, accept placement of indwelling catheter for infusion and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies).
* A positive urine drug screen for cocaine, tetrahydrocannabinol (THC), opiates/opioids, benzodiazepines and amphetamines.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Area under the Concentration-Time Curve (AUC) | 96 hours
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 96 hours
  Maximum Observed Plasma Concentration
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 96 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 96 hours
  Time to Reach Maximum Observed Plasma Concentration
Plasma Decay Half-Life (t1/2) | 96 hours
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Systemic Clearance (CL) | 96 hours
  CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Volume of Distribution at Steady State (Vss) | 96 hours
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Quotient Clinical, Ruddington Fields, Nottingham, United Kingdom

REFERENCES:
- [Derived] Hsyu PH, Pignataro DS, Matschke K. Absolute Bioavailability of Bosutinib in Healthy Subjects From an Open-Label, Randomized, 2-Period Crossover Study. Clin Pharmacol Drug Dev. 2018 May;7(4):373-381. doi: 10.1002/cpdd.396. Epub 2017 Oct 23. PMID 29058816
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1871044&StudyName=Absolute%20Bioavailability%20Of%20Bosutinib